CLINICAL TRIAL: NCT00782353
Title: A Phase 1, Randomized, Double-Blind, Ascending Multiple-Dose Study of the Safety, Tolerability, and Antiviral Activity of ANA598 in Patients With Chronic Hepatitis C Infection
Brief Title: Safety, Tolerability, and Antiviral Activity of ANA598 in Patients With Genotype-1 Chronic HCV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANA598-502
Record Dates: First submitted 2008-10-28; First posted 2008-10-31 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Hepatitis C
Keywords: HCV
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — setrobuvir; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Subjects randomized 8:2 (active:placebo) to receive ANA598 200 mg bid
  Interventions: Drug: ANA598 200 mg bid or placebo
- Cohort 2 (Experimental): Subjects randomized 8:2 (active:placebo) to receive ANA598 400 mg bid
  Interventions: Drug: ANA598 400 mg bid or placebo
- Cohort 3 (Experimental): Subjects randomized 8:2 (active:placebo) to receive ANA598 800 mg bid
  Interventions: Drug: ANA598 800 mg bid or placebo

INTERVENTIONS:
Drug: ANA598 200 mg bid or placebo — ANA598 200 mg bid or placebo
  Arms: Cohort 1
Drug: ANA598 400 mg bid or placebo — ANA598 400 mg bid or placebo
  Arms: Cohort 2
Drug: ANA598 800 mg bid or placebo — ANA598 800 mg bid or placebo
  Arms: Cohort 3

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, and antiviral activity of ANA598 in patients with genotype-1 chronic hepatitis C infection.

DETAILED DESCRIPTION:
The safety, tolerability and antiviral activity of ANA598, administered orally twice daily for 3 days, will be compared to placebo in treatment-naïve subjects chronically infected with HCV genotype 1 infection. Thirty (30) subjects will be randomized to one of three cohorts described above. The ten patients in each cohort will be randomized 8 active: 2 placebo. At least 5 subjects with genotype 1a and 5 subjects with genotype 1b will be enrolled within each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 18 to 65 years
* Documented chronic HCV infection, genotype 1a or 1b
* Treatment-naïve
* BMI = 18 - 35 kg/m2

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Previous treatment for HCV infection
* HIV or HBV positive
* Evidence of cirrhosis on previous liver biopsy or on previous imaging studies
* History of any other known cause of liver disease;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of ascending multiple oral doses of ANA598 administered for 3 days to adult patients with chronic HCV infection and compensated liver disease; | 10 days
The antiviral activity of ANA598, assessed by changes in serum HCV RNA levels | 10 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - United States, Missouri, St Louis, Missouri
  - United States, New York, New York, New York
  - United States, Texas, San Antonio, Texas
- Puerto Rico, Santurce, Santurce, Puerto Rico

REFERENCES:
- [Derived] Mallalieu NL, Rahimy MH, Crowley CA, Appleman JR, Smith PF, Freddo JL. Pharmacokinetics and pharmacodynamics of setrobuvir, an orally administered hepatitis C virus non-nucleoside analogue inhibitor. Clin Ther. 2014 Dec 1;36(12):2047-2063.e3. doi: 10.1016/j.clinthera.2014.10.002. Epub 2014 Nov 4. PMID 25456558